CLINICAL TRIAL: NCT02694133
Title: Efficacy of Telerehabilitation in the Patients With Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Chun-Han Yang, Physical Therapist, Kaohsiung Veterans General Hospital.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS-CT11-06
Record Dates: First submitted 2011-12-27; First posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Aphasia
Keywords: telerehabilitation; aphasia; speech therapy; rehabilitation device; visual action therapy; naming drills
MeSH Terms: conditions — Aphasia; Communication Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aphasia group (Experimental): Aphasia
  Interventions: Procedure: Smart Phone Based Assistive Speech Therapeutic System; Procedure: Mobile phone-based tele rehabilitation program

INTERVENTIONS:
Procedure: Smart Phone Based Assistive Speech Therapeutic System — use the mobile device, which with the camera and speaker, for patients to practice the naming training at home, and assess the speech ability every 2-4weeks by speech therapist via telerehabilitation platform. Concise Chinese Aphasia Test (CCAT) will be used as the assessment tool for evaluation speech ability and functional ability.
Procedure: Mobile phone-based tele rehabilitation program — Mobile phone-based tele rehabilitation program

SUMMARY:
The study will invite 30 patients to join, and they will be arranged in the face to face group and telerehabilitation group randomly.

In the telerehabilitation group, the investigators use the mobile device, which with the camera and speaker, for patients to practice the naming training at home, and assess the speech ability every 2-4weeks by speech therapist via telerehabilitation platform.

Concise Chinese Aphasia Test (CCAT) and ASHA FACS conceptual framework Test will be used as the assessment tool for evaluation speech ability and functional ability.

The investigators expect that patients can improve their speech ability, functional ability, and quality of life via telerehabilitation speech therapy.

And the investigators can establish the standard telerehabilitation speech therapy protocol for aphasia therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as aphasia

Exclusion Criteria:

* poor auditory comprehension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Concise Chinese Aphasia Test | monthly changes within 3 months